Official Title: Assessing Patient Anxiety During Mohs Micrographic Surgery

NCT03756792

IRB Approval Date: 11/28/2020

# **Assessing Patient Anxiety During Mohs Micrographic Surgery**

# Study Fact Sheet Steven R. Feldman, M.D., Ph.D., Principal Investigator

#### INTRODUCTION

You are receiving this document because you have been/will be seen by a dermatologist at Wake Forest Baptist Hospital. We would like to invite you to participate in a research study that will help us better understand the experiences of patients undergoing Mohs Micrographic Surgery in our community.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to learn more about patient's perception of Mohs surgery.

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

100 people at 1 research site will take part in this study.

### WHAT IS INVOLVED IN THE STUDY?

We would like for you to answer a few questions about your level of comfort during the Mohs micrographic surgery. You will be randomized into one of the study groups described below. Randomization means that you are put into a group by chance, much like flipping a coin. You will have an equal chance of being placed into either group. You will be randomly assigned to one of two groups. One group will receive short vignettes about Mohs surgery in addition to standard educational handouts, and the other group will only receive standard educational handouts. You will then be asked to complete a brief survey. This survey includes up to ten questions and will take approximately five minutes to complete. The survey is anonymous; no identifying information will be collected. By completing this survey, you are agreeing to participate in research. The link to the survey with the consent statement can be found here:

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for 1 day.

#### WHAT ARE THE RISKS OF THE STUDY?

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope the information learned from this study will benefit other people in the future. In this study you may or may not benefit from a reduction of anxiety during Mohs surgery.

## WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

It is important that you know that this document is not to tell you to join this study. It is your decision. Your participation is voluntary. While we hope you will consider participating, whether or not you participate in this study will have no effect on your relationship with Wake Forest Baptist Health as a patient.

#### IS PAYMENT AVAILABLE?

You will not be paid for your participation in this study.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

| This is an approved Institutional Review Board (IRB) research study: IRB00054156 at the Wake |
|---|
| Forest University School of Medicine (WFUSM). For questions about the study contact the study |
| investigator, Steven R. Feldman, M.D., Ph.D. at |
| or The Institutional Review Board (IRB) a group of people who |
| review the research to protect your rights. If you have a question about your rights as a research |
| participant, or you would like to discuss problems or concerns, have questions or want to offer |
| input, or you want to obtain additional information, you should contact the Chairman of the IRB |
| . Completion of the survey implies your consent to participate in the study. If |
| you have any further questions about this survey, please do not hesitate to contact our study |
| coordinator Courtney Heron at or Email: |